CLINICAL TRIAL: NCT02918318
Title: A Randomized, Double-blind, Multicenter, Placebo-controlled Study to Evaluate the Efficacy, Safety and Tolerability of Fixed Doses of Intranasal Esketamine in Japanese Subjects With Treatment Resistant Depression
Brief Title: A Study to Evaluate the Efficacy, Safety and Tolerability of Fixed Doses of Intranasal Esketamine in Japanese Participants With Treatment Resistant Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108227; 54135419TRD2005 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2016-09-27; First posted 2016-09-28 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Experimental): Participant will receive 1 spray of placebo to each nostril at 0 minute, 5 minutes and 10 minutes.
  Interventions: Drug: Placebo
- Esketamine 28 milligram (mg) (Experimental): Participant will receive 1 spray of Esketamine to each nostril at 0 minute and placebo at 5 minutes and 10 minutes.
  Interventions: Drug: Intranasal esketamine (28 mg)
- Esketamine 56 mg (Experimental): Participant will receive 1 spray of Esketamine to each nostril at 0 minute, 5 minutes and placebo at 10 minutes.
  Interventions: Drug: Intranasal esketamine (56 mg)
- Esketamine 84 mg (Experimental): Participant will receive 1 spray of Esketamine to each nostril at 0 minute, 5 minutes and 10 minutes.
  Interventions: Drug: Intranasal esketamine (84 mg)

INTERVENTIONS:
Drug: Placebo — Participant will receive 1 spray of placebo to each nostril at 0 minute, 5 minutes and 10 minutes.
  Arms: Placebo
Drug: Intranasal esketamine (28 mg) — Participant will receive 1 spray of Esketamine to each nostril at 0 minute and placebo at 5 minutes and 10 minutes.
  Arms: Esketamine 28 milligram (mg)
Drug: Intranasal esketamine (56 mg) — Participant will receive 1 spray of Esketamine to each nostril at 0 minute, 5 minutes and placebo at 10 minutes.
  Arms: Esketamine 56 mg
Drug: Intranasal esketamine (84 mg) — Participant will receive 1 spray of Esketamine to each nostril at 0 minute, 5 minutes and 10 minutes.
  Arms: Esketamine 84 mg

SUMMARY:
The purpose of this study is to evaluate the efficacy of fixed dosed intranasal esketamine compared to intranasal placebo, as an add-on to an oral antidepressant in Japanese participants with treatment-resistant depression (TRD), in improving depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* At the start of the screening phase, participant must meet the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) diagnostic criteria for single-episode major depressive disorder (MDD) or recurrent major depressive disorder (MDD), without psychotic features, based upon clinical assessment and confirmed by the Mini International Neuropsychiatric Interview (MINI). In the case of single-episode MDD, the participant must be diagnosed with persistent depressive disorder, which meets criteria of major depressive episode for a continuous duration of greater than or equal to (>=)2 years, and the same physician from the site must be examining the participant for >=2 years continuously as a primary care physician of the participant
* The participant's current major depressive episode, depression symptom severity (MADRS total score greater than or equal to [>=] 28 required), and antidepressant treatment response in the current depressive episode, must be confirmed using the SAFER interview
* Participant must be medically stable on the basis of clinical laboratory tests, physical examination, medical history, vital signs (including blood pressure), pulse oximetry, and 12-lead electrocardiogram (ECG) performed in the screening phase
* A woman of childbearing potential must have a negative highly sensitive serum Beta (β) human chorionic gonadotropin [β-hCG] test at the start of the screening phase and a negative urine pregnancy test must be obtained before the first dose of study drug on Day 1 of the double-blind induction phase prior to randomization
* Contraceptive use by men or women should be consistent with local regulations regarding the use of contraceptive methods for participant participating in clinical studies

Exclusion Criteria:

* Participant has received vagal nerve stimulation or has received deep brain stimulation in the current episode of depression
* Participant previously received esketamine or ketamine as treatment for their MDD
* Participant has homicidal ideation/intent, per the investigator's clinical judgment, or has suicidal ideation with some intent to act within 6 months prior to the start of the screening phase
* Participant has a history of moderate or severe substance or alcohol use disorder according to DSM-5 criteria, except nicotine or caffeine, within 6 months before the start of the screening phase
* Participant has a current or past history of seizure disorder (uncomplicated childhood febrile seizures with no sequelae are not exclusionary)

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 202 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (43):
- Japan (43):
  - Akita
  - Fukui-shi
  - Fukuoka
  - Gunma
  - Hachinohe-shi
  - Hachioji-shi
  - Hirakata
  - Hiratsuka-shi
  - Hokkaido
  - Ibaraki
  - Ichikawa
  - Kanzaki-gun
  - Karatsu
  - Kashihara
  - Kawasaki
  - Kita-Azumi
  - Kita-ku
  - Kitakyushu
  - Kobe
  - Kochi
  - Kodaira
  - Komoro-shi
  - Kumamoto
  - Kure
  - Kurume-shi
  - Kyoto
  - Maizuru
  - Morioka
  - Nagakute
  - Nagasaki
  - Okayama
  - Okinawa
  - Osaka
  - Sapporo
  - Setagaya-ku
  - Shibuya-ku
  - Shinjuku
  - Shinjuku-ku
  - Takatsuki-shi
  - Toyoake
  - Ube
  - Yokohama
  - Yonago

REFERENCES:
- [Derived] Ohnishi T, Wakamatsu A, Kobayashi H. Different symptomatic improvement pattern revealed by factor analysis between placebo response and response to Esketamine in treatment resistant depression. Psychiatry Clin Neurosci. 2022 Aug;76(8):377-383. doi: 10.1111/pcn.13379. Epub 2022 Jun 9. PMID 35596932
- [Derived] Takahashi N, Yamada A, Shiraishi A, Shimizu H, Goto R, Tominaga Y. Efficacy and safety of fixed doses of intranasal Esketamine as an add-on therapy to Oral antidepressants in Japanese patients with treatment-resistant depression: a phase 2b randomized clinical study. BMC Psychiatry. 2021 Oct 25;21(1):526. doi: 10.1186/s12888-021-03538-y. PMID 34696742
- See also: A Randomized, Double-blind, Multicenter, Placebo-controlled Study to Evaluate the Efficacy, Safety and Tolerability of Fixed Doses of Intranasal Esketamine in Japanese Subjects With Treatment Resistant Depression — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR108227&attachmentIdentifier=4ef2af53-80a3-47f9-910f-3be69900934c&fileName=54135419TRD2005_(CR108227)_Additional_Results_Data_CH.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Esketamine 28 Milligrams (mg): Double-blind (DB) induction phase: Participants received intranasal esketamine (Esk) 28 mg twice a week add-on to an oral antidepressant (AD) for 4 weeks. Responders (participants who had >=50% reduction from baseline in MADRS total score) at the end of the DB induction phase were eligible to proceed to the posttreatment. DB Follow-up Phase: Participants who did not respond (non-responders) in DB induction phase proceeded to the 4-week DB follow-up and received only oral AD. Posttreatment phase: Participants who were responders at the end of DB induction phase entered in posttreatment phase and received oral AD once daily for up to 24 weeks.
- Esketamine 56 mg: DB induction phase: Participants received intranasal Esk 56 mg twice a week add-on to a AD for 4 weeks. Responders (participants who had >=50% reduction from baseline in MADRS total score) at the end of the DB induction phase were eligible to proceed to the posttreatment. DB Follow-up Phase: Participants who did not respond (non-responders) in DB induction phase proceeded to the 4-week DB follow-up and received only oral AD. Posttreatment phase: Participants who were responders at the end of DB induction phase entered in posttreatment phase and received oral AD once daily for up to 24 weeks.
- Esketamine 84 mg: DB induction phase: Participants received intranasal Esk 84 mg twice a week add-on to AD for 4 weeks. Responders (participants who had >=50% reduction from baseline in MADRS total score) at the end of the DB induction phase were eligible to proceed to the posttreatment. DB Follow-up Phase: Participants who did not respond (non-responders) in DB induction phase proceeded to the 4-week DB follow-up and received only oral AD. Posttreatment phase: Participants who were responders at the end of DB induction phase entered in posttreatment phase and received oral AD once daily for up to 24 weeks.
- Placebo: DB induction phase: Participants received intranasal Esk placebo twice a week add-on to AD for 4 weeks. Responders (participants who had >=50% reduction from baseline in MADRS total score) at the end of the DB induction phase were eligible to proceed to the posttreatment. DB Follow-up Phase: Participants who did not respond (non-responders) in DB induction phase proceeded to the 4-week DB follow-up and received only oral AD. Posttreatment phase: Participants who were responders at the end of DB induction phase entered in posttreatment phase and received oral AD once daily for 24 weeks.
- Esketamine: Flexible Dose: OL induction phase: Responders from the DB induction phase who relapsed in the postreatment phase entered in an open label extension phase and received induction with flexible intransal Esketamine (either 28 mg, 56 mg, or 84 mg) along with oral AD for 4 weeks. OL Follow-up phase: All participants who entered the OL induction phase are followed up in OL follow-up phase for 4 weeks.
Period: Double-blind Induction Phase: 4 Weeks
Arm/Group | Esketamine 28 Milligrams (mg) | Esketamine 56 mg | Esketamine 84 mg | Placebo | Esketamine: Flexible Dose
Started | 41 | 40 | 41 | 80 | 0
Responders | 13 | 11 | 17 | 27 | 0
Completed | 39 | 33 | 39 | 72 | 0
Not Completed | 2 | 7 | 2 | 8 | 0
Not completed — Adverse Event | 1 | 4 | 2 | 3 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0
Not completed — Non-compliance | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 2 | 0 | 1 | 0
Period: Double-blind Follow-up Phase: 4 Weeks
Arm/Group | Esketamine 28 Milligrams (mg) | Esketamine 56 mg | Esketamine 84 mg | Placebo | Esketamine: Flexible Dose
Started | 27 | 28 | 24 | 53 | 0
Completed | 26 | 28 | 23 | 50 | 0
Not Completed | 1 | 0 | 1 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 1 | 0
Period: Posttreatment Phase: Up to 24 Weeks
Arm/Group | Esketamine 28 Milligrams (mg) | Esketamine 56 mg | Esketamine 84 mg | Placebo | Esketamine: Flexible Dose
Started | 13 | 11 | 17 | 27 | 0
Completed | 12 | 8 | 16 | 25 | 0
Not Completed | 1 | 3 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 3 | 1 | 1 | 0
Period: Open Label Treatment Phase: 4 Weeks
Arm/Group | Esketamine 28 Milligrams (mg) | Esketamine 56 mg | Esketamine 84 mg | Placebo | Esketamine: Flexible Dose
Started | 0 | 0 | 0 | 0 | 48
Completed | 0 | 0 | 0 | 0 | 47
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Period: Open Label Follow-up Phase: 4 Weeks
Arm/Group | Esketamine 28 Milligrams (mg) | Esketamine 56 mg | Esketamine 84 mg | Placebo | Esketamine: Flexible Dose
Started | 0 | 0 | 0 | 0 | 48
Completed | 0 | 0 | 0 | 0 | 47
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of intranasal study agent.
Groups:
- Total: Total of all reporting groups
Arm/Group | Esketamine 28 Milligrams (mg) | Esketamine 56 mg | Esketamine 84 mg | Placebo | Total
Number analyzed (Participants) | 41 | 40 | 41 | 80 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (9.97) | 42.5 (8.36) | 41.9 (10.26) | 43.3 (11.4) | 43.4 (10.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 16 | 18 | 39 | 96
  Male | 18 | 24 | 23 | 41 | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 41 | 40 | 41 | 80 | 202
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 41 | 40 | 41 | 80 | 202
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  JAPAN | 41 | 40 | 41 | 80 | 202

OUTCOME MEASURES:

1. Primary Outcome: Double-Blind (DB) Induction Phase: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score up to Day 28
Description: MADRS is clinician-rated scale designed to measure depression severity, and to detect changes due to antidepressant treatment. Scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of symptoms), summed for a total possible score of 0 to 60. Higher scores represent more severe condition. Negative change in score indicates improvement.
Time Frame: Baseline (Day 1) up to Day 28 (DB phase) induction
Population: Full analysis set (FAS [DB]) included all randomized participants who received at least 1 dose of intranasal study agent during the DB induction phase. Here, N (Number of participants analyzed) signifies those participants who were evaluable for this outcome measure (OM).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Esketamine 28 Milligrams (mg) | Esketamine 56 mg | Esketamine 84 mg | Placebo
Number analyzed (Participants) | 39 | 34 | 39 | 72
Units on a scale | -15.2 (13.07) | -14.5 (10.53) | -15.1 (12.21) | -15.3 (11.68)
Statistical Analysis 1: Comparison: Esketamine 28 Milligrams (mg) vs Placebo; Test type: Superiority; p = 0.475, Dunnett adjustment — 1-sided; Difference of Least Squares means = -1.0, 90% CI 2-sided [-5.77 to 3.70], Standard Error of Mean 2.25
Statistical Analysis 2: Comparison: Esketamine 56 mg vs Placebo; Test type: Superiority; p = 0.504, Dunnett adjustment — 1-sided; Difference of Least Squares means = 0.6, 90% CI 2-sided [-4.32 to 5.47], Standard Error of Mean 2.33
Statistical Analysis 3: Comparison: Esketamine 84 mg vs Placebo; Test type: Superiority; p = 0.482, Dunnett adjustment — 1-sided; Difference of Least Squares means = -0.9, 90% CI 2-sided [-5.66 to 3.83], Standard Error of Mean 2.26

2. Secondary Outcome: DB Induction Phase: Percentage of Participants With Response Based on MADRS Total Score
Description: A participant is defined as responder (yes=1 and no=0) at a given time point if the percent improvement from baseline in MADRS is greater than or equal to (>=) 50 percent (%). MADRS is clinician-rated scale designed to measure depression severity, and to detect changes due to antidepressant treatment. Scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of symptoms), summed for a total possible score of 0 to 60. Higher scores represent more severe condition.
Time Frame: Days 2, 8, 15, 22 and 28 (DB induction phase)
Population: FAS (DB) included all randomized participants who received at least 1 dose of intranasal study agent during the DB induction phase. Here 'n' (number analyzed) signifies number of participants who were evaluable for this OM at specified timepoints.
Measure: Number; unit: Percentage of participants
Arm/Group | Esketamine 28 Milligrams (mg) | Esketamine 56 mg | Esketamine 84 mg | Placebo
Number analyzed (Participants) | 41 | 40 | 41 | 80
Percentage of participants
  Day 2: number analyzed (Participants) | 41 | 38 | 40 | 79
  Day 2 | 22.0 | 13.2 | 10.0 | 9.0
  Day 8: number analyzed (Participants) | 41 | 39 | 41 | 79
  Day 8 | 2.4 | 2.6 | 9.8 | 3.8
  Day 15: number analyzed (Participants) | 40 | 36 | 40 | 77
  Day 15 | 17.5 | 8.3 | 15.0 | 18.2
  Day 22: number analyzed (Participants) | 39 | 36 | 39 | 74
  Day 22 | 23.1 | 13.9 | 20.5 | 29.7
  Day 28: number analyzed (Participants) | 39 | 34 | 39 | 72
  Day 28 | 33.3 | 35.3 | 43.6 | 37.5

3. Secondary Outcome: DB Induction Phase: Percentage of Participants With Remission Based on MADRS Total Score
Description: A participant was considered in remission at a given time point if the MADRS total score <=12. MADRS is clinician-rated scale designed to measure depression severity, and to detect changes due to antidepressant treatment. Scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of symptoms), summed for a total possible score of 0 to 60. Higher scores represent more severe condition.
Time Frame: Days 2, 8, 15, 22 and 28 (DB induction phase)
Population: FAS (DB) included all randomized defined as all participants who received at least 1 dose of intranasal study agent during the DB induction phase. Here 'n' (number analyzed) signifies number of participants who were evaluable for this OM at specified timepoints.
Measure: Number; unit: Percentage of participants
Arm/Group | Esketamine 28 Milligrams (mg) | Esketamine 56 mg | Esketamine 84 mg | Placebo
Number analyzed (Participants) | 41 | 40 | 41 | 80
Percentage of participants
  Day 2: number analyzed (Participants) | 41 | 38 | 40 | 78
  Day 2 | 9.8 | 0 | 7.5 | 3.8
  Day 8: number analyzed (Participants) | 41 | 39 | 41 | 79
  Day 8 | 2.4 | 0 | 4.9 | 1.3
  Day 15: number analyzed (Participants) | 40 | 36 | 40 | 77
  Day 15 | 7.5 | 2.8 | 10.0 | 3.9
  Day 22: number analyzed (Participants) | 39 | 36 | 39 | 74
  Day 22 | 10.3 | 5.6 | 7.7 | 14.9
  Day 28: number analyzed (Participants) | 39 | 34 | 39 | 72
  Day 28 | 23.1 | 11.8 | 23.1 | 20.8

4. Secondary Outcome: DB Induction Phase: Percentage of Participants Showing Onset of Clinical Response
Description: A participant was defined as having a clinical response if there was at least 50% improvement from baseline in the MADRS total score with onset by Day 2 that was maintained to Day 28 in DB induction phase. Participants were allowed one excursion (non-response) on Days 8, 15 or 22, provided the score is at least 25% improvement. MADRS is clinician-rated scale designed to measure depression severity, and to detect changes due to antidepressant treatment. Scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of symptoms), summed for a total possible score of 0 to 60. Higher scores represent more severe condition.
Time Frame: Day 2 up to Day 28 (DB induction phase)
Population: FAS (DB) included all randomized participants who received at least 1 dose of intranasal study agent during DB induction phase. Participants with missed assessments or discontinued early were not considered to have onset of clinical response. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this OM.
Measure: Number; unit: Percentage of participants
Arm/Group | Esketamine 28 Milligrams (mg) | Esketamine 56 mg | Esketamine 84 mg | Placebo
Number analyzed (Participants) | 41 | 39 | 41 | 79
Percentage of participants
  Onset of clinical response: Yes | 2.4 | 2.6 | 7.3 | 6.3
  Onset of clinical response: No | 97.6 | 97.4 | 92.7 | 93.7

5. Secondary Outcome: DB Induction Phase: Change From Baseline in Clinical Global Impression - Severity (CGI-S) Total Score up to Day 28
Description: CGI-S provides measure of severity of participant's illness including participant's history, psychosocial circumstances, symptoms, behavior and impact of symptoms on ability to function. CGI-S evaluates severity of psychopathology on scale of 0 to 7. Considering total clinical experience, participant is assessed on severity of mental illness according to: 0=not assessed; 1=normal (not at all ill); 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among most extremely ill patients. Values of 0 (not assessed) were excluded from analysis. CGI-S permits global evaluation of participant's condition at given time.
Time Frame: Baseline (Day 1) up to Day 28 (DB induction pahse)
Population: FAS (DB) included all randomized participants who received at least 1 dose of intranasal study agent during the DB induction phase. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this OM.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Esketamine 28 Milligrams (mg) | Esketamine 56 mg | Esketamine 84 mg | Placebo
Number analyzed (Participants) | 39 | 33 | 39 | 72
Units on a scale | -1.0 [-5 to 1] | -1.0 [-3 to 0] | -1.0 [-5 to 0] | -1.0 [-4 to 1]

6. Secondary Outcome: DB Induction Phase: Change From Baseline in Generalized Anxiety Disorder 7-Item Scale (GAD-7) up to Day 28
Description: GAD-7 was a brief and validated 7-item self-report assessment of overall anxiety. Participants respond to each item using a 4-point scale with response categories of 0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day. Item responses are summed to yield a total score with a range of 0 to 21, where higher scores indicate more anxiety. The recall period is 2 weeks. The severity of the GAD-7 is categorized as follows: None (0-4), Mild (5-9), Moderate (10-14) and Severe (15 -21).
Time Frame: Baseline (Day 1) up to Day 28 (DB induction phase)
Population: FAS included all randomized participants who received at least 1 dose of intranasal study agent during the DB induction phase. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this OM.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Esketamine 28 Milligrams (mg) | Esketamine 56 mg | Esketamine 84 mg | Placebo
Number analyzed (Participants) | 39 | 35 | 39 | 73
Units on a scale | -8.2 (4.94) | -7.8 (5.05) | -8.1 (5.67) | -7.7 (5.05)

7. Secondary Outcome: DB Induction Phase: Change From Baseline in Sheehan Disability Scale (SDS) Total Score up to Day 28
Description: SDS is a participant-reported outcome measure and 5 item questionnaire used for assessment of functional impairment and associated disability. First three items assess disruption of 1 work/school, 2 social life, 3 family life/home responsibilities using a 0(no impairment)-10 (most severe impairment). Score for first 3 items are summed to create total score of 0-30 where higher score indicates greater impairment and a negative change in score indicates improvement. It also has one item on days lost from school or work and one item on days when under productive.
Time Frame: Baseline (Day 1) to Day 28 (DB induction phase)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Esketamine 28 Milligrams (mg) | Esketamine 56 mg | Esketamine 84 mg | Placebo
Number analyzed (Participants) | 30 | 29 | 31 | 53
Units on a scale | -8.6 (8.68) | -7.9 (7.94) | -9.5 (8.93) | -7.0 (7.39)

8. Secondary Outcome: Posttreatment Phase: Time to Relapse in Participants With Remission (MADRS Total Score <=12)
Description: Time to relapse in participants with remission at the end of the double-blind phase was defined as the time between induction phase and the first documentation of a relapse event during the posttreatment phase. Relapse was defined as any of the following: 1) MADRS total score >= 22 for 2 consecutive assessments. The date of the second MADRS assessment was used for the date of relapse; 2) Hospitalization for worsening depression or any other clinically relevant event determined per clinical judgment to be suggestive of relapse of depressive illness like suicide attempt, completed suicide, or hospitalization for suicide prevention. If hospitalized for any of these events, start date of hospitalization was used as relapse date. If participant was not hospitalized, event date was used. 3) If both relapse criteria were met, earlier date was defined as date of relapse. Remission was defined as MADRS total score <=12.
Time Frame: From EndPoint (last post baseline assessment value during the DB induction phase [up to Day 28]) up to 24 weeks (posttreatment phase)
Population: Population included participants with remit at the end of DB.
Measure: Median (90% Confidence Interval); unit: Days
Arm/Group | Esketamine 28 Milligrams (mg) | Esketamine 56 mg | Esketamine 84 mg | Placebo
Number analyzed (Participants) | 9 | 4 | 9 | 15
Days | 34.0 [26.0 to NA] — Upper limit of 90 % confidence internal was not estimable due to insufficient number of participants with events. | 52.0 [20.0 to 80.0] | 37.0 [19.0 to 71.0] | 30.0 [22.0 to 50.0]

9. Secondary Outcome: Posttreatment Phase: Time to Relapse in Participants With Response (>=50% Reduction From Baseline in MADRS Total Score) But Who Are Not in Remission
Description: Time to relapse in participants with response (>=50% reduction from baseline in MADRS total score) but who are not in remission was reported. Relapse is defined as any of the following: 1) MADRS total score >= 22 for 2 consecutive assessments. The date of the second MADRS assessment was used for the date of relapse. 2)Hospitalization for worsening depression or any other clinically relevant event determined per clinical judgment to be suggestive of relapse of depressive illness like suicide attempt, completed suicide, or hospitalization for suicide prevention. If hospitalized for any of these events, start date of hospitalization was used as relapse date. If participant was not hospitalized, event date was used. 3) If both relapse criteria were met, earlier date was defined as date of relapse. Remission was defined as MADRS total score <=12.
Time Frame: as for outcome 8
Population: Population included participants with response (not remit) at the end of DB.
Measure: Median (90% Confidence Interval); unit: Days
Arm/Group | Esketamine 28 Milligrams (mg) | Esketamine 56 mg | Esketamine 84 mg | Placebo
Number analyzed (Participants) | 13 | 11 | 17 | 27
Days | 32.0 [13.0 to 44.0] | 26.0 [9.0 to 121.0] | 79.5 [16.0 to 108.0] | 91.0 [22.0 to NA] — Upper limit of 90 % confidence internal was not estimable due to insufficient number of participants with events.

10. Secondary Outcome: Posttreatment Phase: Change From Baseline in Sheehan Disability Scale (SDS) Total Score at Weeks 2, 4, 6, 8, 12, 16, 20 and 24
Description: SDS is a participant-reported outcome measure and is a 5-item questionnaire which has been widely used and accepted for assessment of functional impairment and associated disability. The first three items assess disruption of (1) work/school, (2) social life, and (3) family life/home responsibilities using a 0-10 rating scale. The score for the first three items are summed to create a total score of 0-30, where a higher score indicates greater impairment. It also has one item on days lost from school or work and one item on days when under productive. FAS (responders): All randomized participants who received at least 1 dose of intranasal study medication during DB induction phase and who were responders at the end of DB induction phase and entered posttreatment phase
Time Frame: Baseline (DB induction phase), Weeks 2, 4, 6, 8, 12, 16, 20 and 24 (posttreatment phase)
Population: Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this OM. Here, 'n' (number analyzed) signifies number of participants who were evaluable for this OM at specified timepoints.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Esketamine 28 Milligrams (mg) | Esketamine 56 mg | Esketamine 84 mg | Placebo
Number analyzed (Participants) | 8 | 10 | 13 | 18
Units on a scale
  Week 2 | -14.6 (7.82) | -8.1 (6.15) | -13.1 (7.65) | -11.2 (6.83)
  Week 4: number analyzed (Participants) | 8 | 7 | 10 | 13
  Week 4 | -12.9 (5.69) | -8.3 (2.75) | -13.6 (7.34) | -9.8 (5.84)
  Week 6: number analyzed (Participants) | 3 | 3 | 8 | 9
  Week 6 | -17.7 (8.50) | -11.0 (3.61) | -14.6 (5.53) | -12.0 (4.39)
  Week 8: number analyzed (Participants) | 3 | 3 | 6 | 7
  Week 8 | -12.0 (14.42) | -13.3 (1.53) | -15.3 (7.15) | -11.4 (6.02)
  Week 12: number analyzed (Participants) | 2 | 3 | 4 | 6
  Week 12 | -20.5 (3.54) | -13.0 (7.21) | -18.3 (7.76) | -14.8 (4.88)
  Week 16: number analyzed (Participants) | 2 | 2 | 2 | 4
  Week 16 | -21.5 (6.36) | -17.5 (0.71) | -12.5 (21.92) | -15.8 (1.89)
  Week 20: number analyzed (Participants) | 2 | 1 | 1 | 4
  Week 20 | -22.0 (7.07) | -18.0 | -28.0 | -14.0 (3.65)
  Week 24: number analyzed (Participants) | 2 | 1 | 1 | 4
  Week 24 | -21.5 (4.95) | -16.0 | -28.0 | -14.8 (3.59)

11. Secondary Outcome: OL Induction Phase: Percentage of Participants With Remission Based on MADRS Total Score
Description: as for outcome 3
Time Frame: Days 8, 15, 22 and 28 (OL induction phase)
Population: FAS (OL) included all randomized participants who received at least 1 dose of intranasal study agent during the OL induction phase. Here 'n' (Number analyzed) signifies number of participants who were evaluable for this OM at specified timepoints.
Measure: Number; unit: Percentage of participants
Arm/Group | Esketamine: Flexible Dose
Number analyzed (Participants) | 48
Percentage of participants
  Day 8 | 14.6
  Day 15: number analyzed (Participants) | 47
  Day 15 | 23.4
  Day 22: number analyzed (Participants) | 47
  Day 22 | 31.9
  Day 28: number analyzed (Participants) | 47
  Day 28 | 42.6

12. Secondary Outcome: OL Induction Phase: Change From Baseline (Prior to the First Dose of OL Induction Phase) in MADRS Total Score up to Endpoint OL Induction Phase (Last Post Baseline Assessment Value During the OL Induction Phase [OL: up to Day 28])
Description: MADRS is clinician-rated scale designed to measure depression severity, and to detect changes due to antidepressant treatment. Scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of symptoms), summed for a total possible score of 0 to 60. Higher scores represent more severe condition.
Time Frame: Baseline (Prior to first Dose of OL induction phase on Day 1) up to endpoint of OL induction phase (last post baseline assessment value during OL induction phase [OL: up to Day 28])
Population: FAS (OL) included all participants who received at least 1 dose of intranasal study agent during the OL induction phase.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Esketamine: Flexible Dose
Number analyzed (Participants) | 48
Units on a scale
  Baseline | 16.1 (9.47)
  Change from baseline | -14.5 (11.06)

13. Secondary Outcome: OL Induction Phase: Percentage of Participants With Severity of Psychopathology on the CGI-S Scale
Description: CGI-S provides measure of severity of participant's illness including participant's history, psychosocial circumstances, symptoms, behavior and impact of symptoms on ability to function. CGI-S evaluates severity of psychopathology on scale of 0 to 7. Considering total clinical experience, participant is assessed on severity of mental illness according to: 0=not assessed; 1=normal (not at all ill); 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among most extremely ill patients. CGI-S permits global evaluation of participant's condition at given time.
Time Frame: Baseline (Prior to first dose of OL induction phase on Day 1), endpoint of OL induction phase (last post baseline assessment value during the OL induction phase [OL: up to Day 28])
Population: FAS (OL) included all participants who received at least 1 dose of intranasal study agent during the OL induction phase.
Measure: Number; unit: Percentage of participants
Arm/Group | Esketamine: Flexible Dose
Number analyzed (Participants) | 48
Percentage of participants
  Normal, not at all ill:Baseline | 0
  Normal, not at all ill:Endpoint | 14.6
  Borderline mentally ill:Baseline | 0
  Borderline mentally ill:Endpoint | 16.7
  Mildly ill:Baseline | 4.2
  Mildly ill:Endpoint | 43.8
  Moderately ill:Baseline | 75.0
  Moderately ill:Endpoint | 20.8
  Markedly ill:Baseline | 14.6
  Markedly ill:Endpoint | 4.2
  Severely ill:Baseline | 4.2
  Severely ill:Endpoint | 0
  Among the most extremely ill patients:Baseline | 2.1
  Among the most extremely ill patients:Endpoint | 0

ADVERSE EVENTS:
Time Frame: Up to 42 weeks
Description: There was 1 participant who was randomized to the Esk 84 mg group but was dosed Esk 56 mg on Days 1 and 4, and Esk 28 mg on Day 8, then withdrew due to an adverse event on Day 11. This participant was summarized under the Esk 56 mg group for safety analyses.
Groups:
- Double Blind (DB): Esketamine 28 mg: Participants received intranasal esketamine 28 mg twice a week add-on to an oral antidepressant (AD) for 4 weeks. Analysis was performed on safety analysis set- all randomized participants who received at least 1 dose of Esk during DB induction phase.
- DB: Esketamine 56 mg: Participants received intranasal esketamine 56 mg twice a week add-on to an oral AD for 4 weeks. Analysis was performed on safety analysis set- all randomized participants who received at least 1 dose of Esk DB induction phase.
- DB: Esketamine 84 mg: Participants received intranasal esketamine 84 mg twice a week add-on to an oral AD for 4 weeks. Analysis was performed on safety analysis set- all randomized participants who received at least 1 dose of Esk during DB induction phase.
- DB: Placebo: Participants received intranasal placebo twice a week add-on to an oral AD for 4 weeks. Analysis was performed on safety analysis set- all randomized participants who received dose of internasal placebo during DB induction phase.
- DB Follow Up (FU): Esketamine 28 mg: Participants who were non responders at the end of DB induction phase and entered the DB follow-up phase received only oral AD for 4 weeks. Analysis was performed on follow-up analysis set- all participants who entered the follow-up phase and were evaluated for the safety.
- DB FU: Esketamine 56 mg; DB FU: Esketamine 84 mg; DB FU: Placebo: Participants who were non responders at the end of DB induction phase and entered the DB follow-up phase received only oral AD in the DB FU phase. Analysis was performed on follow-up analysis set- all participants who entered the follow-up phase and were evaluated for the safety.
- Post-Treatment (PT) Phase: Esketamine 28 mg; PT Phase: Esketamine 56 mg; PT Phase: Placebo: Participants who were responders at the end of DB induction phase and entered in the PT phase received only oral AD in the PT phase. Analysis was performed on safety analysis set- All participants who received at least 1 dose of oral AD during PT phase.
- PT Phase: Esketamine 84 mg: Participants who were responders at the end of DB induction phase and entered in the PT phase received only an oral AD in the PT phase. Analysis was performed on safety analysis set- All participants who received at least 1 dose of oral AD during PT phase.
- Open-Label (OL): Flexible Esketamine: Participants received flexible esketamine add-on to an oral AD during OL induction phase for 4 weeks. Analysis was performed on safety analysis set- All participants who received at least 1 dose of flexible Esk during OL induction phase.
- OL FU: Flexible Esketamine: Participants who received flexible esketamine add-on to an oral AD during OL induction phase were followed for 4 weeks in OL FU phase. Analysis was performed on follow-up analysis set- all participants who entered the OL follow-up phase and were evaluated for the safety.
Arm/Group | Double Blind (DB): Esketamine 28 mg | DB: Esketamine 56 mg | DB: Esketamine 84 mg | DB: Placebo | DB Follow Up (FU): Esketamine 28 mg | DB FU: Esketamine 56 mg | DB FU: Esketamine 84 mg | DB FU: Placebo | Post-Treatment (PT) Phase: Esketamine 28 mg | PT Phase: Esketamine 56 mg | PT Phase: Esketamine 84 mg | PT Phase: Placebo | Open-Label (OL): Flexible Esketamine | OL FU: Flexible Esketamine
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/41 | 0/40 | 0/80 | 0/27 | 0/29 | 0/23 | 0/53 | 0/13 | 0/11 | 0/17 | 0/27 | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 1/41 | 0/41 | 1/40 | 1/80 | 0/27 | 0/29 | 1/23 | 2/53 | 0/13 | 0/11 | 0/17 | 0/27 | 1/48 | 2/48
Other Adverse Events (participants affected / at risk) | 33/41 | 39/41 | 39/40 | 34/80 | 3/27 | 3/29 | 3/23 | 7/53 | 6/13 | 4/11 | 6/17 | 7/27 | 47/48 | 3/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind (DB): Esketamine 28 mg (N=41) | DB: Esketamine 56 mg (N=41) | DB: Esketamine 84 mg (N=40) | DB: Placebo (N=80) | DB Follow Up (FU): Esketamine 28 mg (N=27) | DB FU: Esketamine 56 mg (N=29) | DB FU: Esketamine 84 mg (N=23) | DB FU: Placebo (N=53) | Post-Treatment (PT) Phase: Esketamine 28 mg (N=13) | PT Phase: Esketamine 56 mg (N=11) | PT Phase: Esketamine 84 mg (N=17) | PT Phase: Placebo (N=27) | Open-Label (OL): Flexible Esketamine (N=48) | OL FU: Flexible Esketamine (N=48)
Atrioventricular Block Second Degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebral Disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicide Attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind (DB): Esketamine 28 mg (N=41) | DB: Esketamine 56 mg (N=41) | DB: Esketamine 84 mg (N=40) | DB: Placebo (N=80) | DB Follow Up (FU): Esketamine 28 mg (N=27) | DB FU: Esketamine 56 mg (N=29) | DB FU: Esketamine 84 mg (N=23) | DB FU: Placebo (N=53) | Post-Treatment (PT) Phase: Esketamine 28 mg (N=13) | PT Phase: Esketamine 56 mg (N=11) | PT Phase: Esketamine 84 mg (N=17) | PT Phase: Placebo (N=27) | Open-Label (OL): Flexible Esketamine (N=48) | OL FU: Flexible Esketamine (N=48)
Palpitations (Cardiac disorders) | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hyperacusis (Ear and labyrinth disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 4 | 7 | 8 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0
Conjunctivitis Allergic (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry Eye (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Visual Impairment (Eye disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 2 | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypoaesthesia Oral (Gastrointestinal disorders) | 3 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Nausea (Gastrointestinal disorders) | 7 | 7 | 8 | 7 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 12 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 4 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Asthenia (General disorders) | 2 | 7 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Feeling Drunk (General disorders) | 1 | 5 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0
Malaise (General disorders) | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Thirst (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 3 | 2 | 1 | 1 | 3 | 2 | 2 | 2 | 3 | 2 | 2
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood Pressure Diastolic Increased (Investigations) | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Pressure Increased (Investigations) | 12 | 19 | 19 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24 | 0
Respiratory Rate Decreased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight Increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 11 | 18 | 15 | 5 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 21 | 0
Dizziness Postural (Nervous system disorders) | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Dyslalia (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 6 | 5 | 4 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 8 | 0
Hypoaesthesia (Nervous system disorders) | 7 | 8 | 5 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 1
Hypotonia (Nervous system disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mental Impairment (Nervous system disorders) | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Sedation (Nervous system disorders) | 1 | 4 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0
Somnolence (Nervous system disorders) | 10 | 13 | 11 | 14 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 11 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Depersonalisation/Derealisation Disorder (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Dissociation (Psychiatric disorders) | 14 | 10 | 22 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 31 | 0
Euphoric Mood (Psychiatric disorders) | 0 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Hallucination (Psychiatric disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Albuminuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Esk has transient dissociative effects that are difficult to blind, these specific events could have biased clinical staff who observed treatment sessions. To ensure an unbiased efficacy evaluation, remote, blinded MADRS raters were used.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2018-12-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT02918318/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/18/NCT02918318/SAP_001.pdf